CLINICAL TRIAL: NCT05958537
Title: Use of High Flow Nasal Oxygen Cannula in Transcatheter Aortic Valve Replacement Procedures. Impact on Respiratory Complications and Biomarkers
Brief Title: High Flow Nasal Oxygen Cannula in Transcatheter Aortic Valve Replacement: Complications and Biomarkers
Acronym: HIGH-OXY-TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2022/1095
Record Dates: First submitted 2023-06-29; First posted 2023-07-24 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2023-06

CONDITIONS: Aortic Stenosis; Sedation Complication
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): In the intervention group, 50 L/min with 0.6 FiO2 will be administered through a high-flow nasal cannula.
  Interventions: Device: High flow nasal oxygen
- Control (No Intervention): In the control group, oxygen therapy will also be administered in all cases, using the usual procedure: oxygen therapy through a conventional nasal cannula and at a flow of 5 L/min

INTERVENTIONS:
Device: High flow nasal oxygen — Use of High-flow nasal oxygen at 60% 50 L/min.
  Arms: Intervention

SUMMARY:
Background Transcatheter aortic valve replacement is a risky procedure, performed in patients that can also be considered at risk of developing complications. The use of HFNO could be justified in this context and could improve the results and safety of these procedures. The use of HFNO during sedation for TAVR could increase oxygen content and minimise hypercapnia, which occurs frequently. This may have 2 potential benefits: one in terms of facilitating the patient's tolerance to anaesthetic sedation; and the other to optimise oxygen delivery to organs such as the brain, kidneys, and myocardium.

Primary aim The number of oxygen desaturation episodes. An oxygen desaturation episode is defined as any episode of Sp02 <93% for more than 10 seconds.

Method A single-center prospective randomised controlled clinical trial with 132 individuals comparing the use of High Flow Nasal oxygen (intervention group) with the conventional standard of care oxygenation with nasal cannula standard oxygenation (control group) of patients undergoing sedation for transfemoral TAVR. The randomisation process will be carried out with a 1:1 assignment, using the RedCap Clínic tool for this purpose. Both groups will be treated at the same centre and by the same interventional cardiology and anaesthesia team. Sedation regime will be based on Target controlled infusion (TCI) with propofol and remifentanil. Local anaesthesia will be infiltrated by interventional cardiologist prior obtaining femoral vascular access. 50 L/min with 0.6% FiO2 will be administered through a high-flow nasal cannula in the intervention group. In the control group, oxygen therapy will also be administered in all cases, using the usual procedure: oxygen therapy through a conventional nasal cannula and at a flow of 5 L/min.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years of age undergoing transfemoral TAVR procedure under local anaesthesia and sedation consenting to participate in the study

Exclusion Criteria:

* <18 years and/or refusal to give informed consent for participation General anaesthesia required to perform complex cases of TAVR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The number of oxygen desaturation episodes | up to 24 hours
  An oxygen desaturation episode is defined as any episode of Sp02 <93% more than 10 seconds
The number of patients with at least 1 desaturation episode | up to 24 hours
  An oxygen desaturation episode is defined as any episode of Sp02 <93% more than 10 seconds

SECONDARY OUTCOMES:
Hypoxia | At placing the arterial catheter moment (baseline), and 45 minutes after the start of sedation
  PO2
Hipercapnia | At placing the arterial catheter moment (baseline), and 45 minutes after the start of sedation
  PaCO2
Trends in plasmatic enolase neurospecific | the day before the procedure (baseline), 45 minutes, and 8 hours after the start of sedation.
  Study of plasmatic biomarkers of ischaemic damage in brain with Enolase neurospecific
Trends in plasmatic Biomarkers of kidney injury | the day before the procedure (baseline), 45 minutes, and 8 hours after the start of sedation.
  Study of plasmatic biomarkers of ischaemic damage in kidney with creatinine
Trends in plasmatic Biomarkers of myocardial injury | the day before the procedure (baseline), 45 minutes, and 8 hours after the start of sedation.
  Study of plasmatic biomarkers of ischaemic damage in myocardium with troponin and pro-BNP
Respiratory depression | During the TAVI procedure
  Number of respiratory depression episodes requiring manual ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No